CLINICAL TRIAL: NCT00619736
Title: Ascending Single Dose Study of the Safety, Tolerability and Pharmacokinetics of NSA-789 Administered Orally to Healthy Japanese Male Subjects
Brief Title: Study Evaluating the Safety, Tolerability and Pharmacokinetics of NSA-789 in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 3230A1-1001
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NSA-789 (Experimental)
  Interventions: Drug: NSA-789
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NSA-789
  Arms: NSA-789
Other: Placebo
  Arms: Placebo

SUMMARY:
This study will provide an initial assessment of the safety, tolerability and pharmacokinetics (PK) of NSA-789 after administration of ascending single oral doses to healthy Japanese male subjects. This is a randomized, double-blind, placebo-controlled, inpatient, sequential-group study conducted under fasting conditions at a single investigational site. Each subject will participate in only 1 dose group and will receive only 1 dose of test article.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 20 to 45 years inclusive at screening.
* Healthy as determined by the investigator on the basis of screening evaluations.

Exclusion Criteria:

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* Use of any investigational drug within 90 days before study day 1 or prescription drug within 30 days before study day 1
* Any clinically important deviation from normal limits in physical examination, vital signs, 12-lead electrocardiograms (ECGs), or clinical laboratory test results.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 3 months

SECONDARY OUTCOMES:
Pharmacokinetics | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer